CLINICAL TRIAL: NCT00742807
Title: Pain Evaluation During Follicle Aspiration: Comparison of Two Sedation Protocols
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No investigator to follow-up
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/291
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pain
Keywords: sensation; relief; during; surgery
MeSH Terms: conditions — Pain | interventions — Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Administration of low dose of alfentanil hydrochloride before paracervical block
  Interventions: Drug: Low dose of alfentanil hydrochloride
- 2 (Active Comparator): Administration of alfentanil hydrochloride dose after paracervical block
  Interventions: Drug: Normal dose of alfentanil hydrochloride

INTERVENTIONS:
Drug: Low dose of alfentanil hydrochloride — Administration of low dose alfentanil hydrochloride before paracervical block
  Arms: 1
Drug: Normal dose of alfentanil hydrochloride — Normal dose of alfentanil hydrochloride is administered after paracervical block
  Arms: 2

SUMMARY:
Giving infiltration analgesia around the neck of the womb (= paracervical block, PCB) is frequently experienced as a painful procedure by women undergoing follicle aspiration. Two sedation protocols, where in the one protocol a low dose of alfentanil hydrochloride is already administered before the PCB, will be compared with each other and pain relief measured using the 'Visual Analogue Scale' and the 'Short-Form McGill Questionnaire'

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and female infertility patients
* Between 18 and 43 years of age

Exclusion Criteria:

* Patients with a known allergy to alfentanil hydrochloride or comparable drugs (morphine, cocaine)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain relief | During and immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dumortier, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Website of the Ghent University Hospital — http://www.uzgent.be